CLINICAL TRIAL: NCT04291703
Title: Low Dose Antithymocyte Globulin (ATG) to Delay or Prevent Progression to Stage 3 T1D
Brief Title: STOP-T1D Low-Dose (ATG)
Acronym: TN28
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated early due to low enrollment and lack of feasibility to meet target enrollment.
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: TrialNet TN28; UC4DK117009-01 (NIH)
Record Dates: First submitted 2020-02-26; First posted 2020-03-02 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: TrialNet; T1D
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Antilymphocyte Serum; thymoglobulin

STUDY DESIGN:
Intervention Model Description: Eligible study participants will be randomized in a 2:1 allocation to either ATG vs. placebo treatment arms by the TrialNet Coordinating Center at the baseline visit once eligibility has been confirmed. Randomization will be conducted using block randomization with variable block sizes with stratification on TrialNet study site and age group (< 12 years old vs. 12 years old or older). Subjects will be assigned a study randomization number corresponding to the treatment group assignment.
Who Masked: Participant, Care Provider, Investigator
Masking Description: The randomization method will be stratified by TrialNet study site. The participants will not be informed regarding the intervention assignment until the end of the study. The investigator and clinic personnel will also be masked as to study assignment. Laboratories performing assays for this protocol will be masked as to the identity of biological material to be studied.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Antithymocyte globulin (ATG) (Experimental): Antithymocyte globulin (ATG) will be intravenously administered over two days, with a total of 2 infusion periods. The first infusion is given at baseline visit (day 1), the second is given the next day at baseline visit (day 2). Body weight at baseline (Day 0- admission for the ATG/placebo infusion) will be used in calculating the doses for all infusions. The first dose (0.5mg/kg) will be infused over a minimum of 4 hours, and the second dose (2mg/kg) over a minimum of 4 hours with a maximum infusion time for each infusion of 10 hours. The second dose should be given no less than 12 and no more than 30 hours from the start of the first infusion. The final prepared product is to be labeled to protect the blind. Infusions may be administered either in a hospital or outpatient setting at the investigator's or institutions discretion.
  Interventions: Drug: Antithymocyte Globulin
- Placebo (Placebo Comparator): 0.9% Sodium Chloride Injection USP ("Normal" saline) is to be dispensed as the placebo for this study. The placebo is to be prepared dispensing an infusion bag of 0.9% Sodium Chloride Injection USP ("Normal" saline) with no additives (no ATG, no premedications) and label the product to protect the blind. The placebo will also be administered over a minimum of 4 hours for the first and second doses with a maximum infusion time of 10 hours. The second dose of the placebo arm should be given no less than 12 and no more than 30 hours from the start of the first infusion. Infusions may be administered either in a hospital or outpatient setting at the investigator's or institutions discretion.
  Interventions: Drug: Placebo (for ATG)

INTERVENTIONS:
Drug: Antithymocyte Globulin — Thymoglobulin
  Other Names: Thymoglobulin
  Arms: Antithymocyte globulin (ATG)
Drug: Placebo (for ATG) — Normal Saline administered by IV infusion to mimic ATG
  Arms: Placebo

SUMMARY:
A multi-center, placebo-controlled, double blind, 2:1 randomized control clinical trial testing low-dose ATG vs. placebo in subjects with a 2 year 50% risk of progression to stage 3 T1D.

DETAILED DESCRIPTION:
This study has an enrollment period of 4 years and once the enrollment phase has concluded, an additional two years of follow-up visits will be conducted for all participants. Participants enrolled in the first year of the study can expect to complete follow-up visits for approximately four additional years if progression to stage 3 (Type 1 Diabetes Onset) does not occur. Participant follow-up visits after the treatment phase of the study includes general assessments (medical history, physical exam, medications and adverse events) and laboratory assessments to determine current health status and glucose tolerance.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to provide informed consent or have a parent or legal guardian provide informed consent when the subject is <18 years of age.
2. Age greater than or equal to 6 and < 35 years
3. At least two or more diabetes-related biochemical autoantibodies (mIAA, GADA, ICA, IA-2A, ZnT8A) present on the same sample. In the absence of other antibodies, ICA and GADA positivity alone will not suffice for eligibility in this trial.
4. Weight greater than the 5th percentile for age and sex.
5. BMI < 95th and > 5th percentile for age for those under age 18 years and < 30 and > 15 for adults (≥ 18)
6. ADA Stage 2 criteria* AND at least one of the following high-risk markers (occurring at the same visit) within 7 weeks (52 days) of randomization, defined below (for defining a 2-year 50% risk for progression to Stage 3 T1D):

   a. HbA1c ≥ 5.7 and <6.5% b. Index60 ≥ 1.4 i. Index60 = 0.3695 × (log fasting C-peptide [ng/mL]) + 0.0165 × 60-min glucose (mg/dL) - 0.3644 × 60-min C-peptide (ng/mL) c. DPTRS ≥ 7.4 DPTRS = (1.57 x log BMI) - (0.06 x age) + (0.81 x glucose sum from 30 to 120 min/100) - (0.85 x C-peptide sum from 30 to 120 min/10) + (0.48 x log fasting C-peptide)

   *Dysglycemia is defined as 2-hr glucose ≥ 140 and <200 mg/dL or fasting glucose ≥ 110 and <126 or 30, 60, or 90 minute glucose ≥ 200 mg/dL from OGTT
7. All subjects must be CMV and EBV PCR negative within 30 days of randomization and may not have had signs or symptoms of a CMV or EBV-compatible illness lasting longer than 7 days within 30 days of randomization
8. Seated blood pressure less than 130/80 mmHg for participants ≥ 18 years. For participants < 18 years seated blood pressure less than 95th percentile for age, sex and height.
9. Be at least 4 weeks from last live immunization
10. Participants are required to receive non-live influenza vaccination at least 2 weeks prior to randomization when vaccine for the current or upcoming flu season is available.
11. Participants must also have a negative COVID-19 test within 7 days of the first day of treatment if otherwise eligible
12. Willingness to comply with study directed social distancing and protection from SARS-Cov-2 infection.
13. Be willing to forgo vaccines (other than killed influenza) during the 3 months after study drug treatment period (Days 0 and 1)
14. Be up to date on all recommended vaccinations based on age of subject*
15. With the exception of stage 2 T1D, subjects must be healthy, as defined by absence of any other untreated diagnoses that the protocol committee deems to be a potential confounder.
16. If a female participant with reproductive potential, willing to avoid pregnancy (abstinence or adequate contraceptive method) through the completion of the study infusions and up to 3 months after study drug administration and undergo pregnancy testing prior to each study visit.
17. Must be residing or have accommodations within 1 hour of the infusion site during the two days of study drug infusions and must be within 1 hour of a medical care facility for 1 day after completion of infusion 2.
18. Participants must live in a location with rapid access to emergency medical services.

    * Adult participants must be fully immunized. Pediatric participants who have not completed their primary vaccination schedule must receive all vaccinations allowable per the national/country-specific immunization guidelines for their current age prior to study drug delivery. Any remaining vaccinations should be given and continue per the schedule at least 3 months after study drug is administered. For COVID-19 vaccination, all participants will be strongly encouraged to be up-to-date with COVID-19 vaccine(s) as indicated by country-specific guidelines at least 2 weeks prior to randomization.

Exclusion Criteria:

1. Immunodeficiency or clinically significant chronic lymphopenia: (Leukopenia (< 3,000 leukocytes /μL), neutropenia (<1,500 neutrophils/μL), lymphopenia (<800 lymphocytes/μL), thrombocytopenia (<100,000 platelets/μL).
2. Hemoglobin less than 13.5 g/dL for adult men and less than 12 g/dL for adult females and less than 11 g/dL for participants under age 18
3. Active signs or symptoms of acute infection at the time of randomization including SARS-Cov-2.
4. Uncontrolled autoimmune thyroid disease and/or celiac disease (participants must be well controlled for the previous 6 months).
5. Evidence of prior or current tuberculosis infection as assessed interferon gamma release assay (QuantiFERON).
6. Currently pregnant or lactating or anticipate getting pregnant within the study period.
7. Require use of other immunosuppressive agents including chronic use of systemic steroids.
8. Evidence of current or past HIV or Hepatitis B or current Hepatitis C infection.
9. Any complicating medical issues or abnormal clinical laboratory results that may interfere with study conduct, or cause increased risk to include pre-existing cardiac disease, COPD, sickle cell disease, neurological disease, or blood count abnormalities.
10. A history of malignancies other than of skin.
11. Evidence of liver dysfunction with AST or ALT outside of the reference range.
12. Evidence of renal dysfunction with creatinine outside of the reference range.
13. Increased bilirubin (total and direct) outside of the normal limit (Participants with documentation of Gilbert's Disease permitted).
14. Vaccination with a live virus within the last 4 weeks.
15. Current or ongoing use of non-insulin pharmaceuticals that affect glycemic control within 7 days of screening
16. Prior treatment with Teplizumab (either in a previous clinical trial or clinically).
17. Has participated in a clinical trial for diabetes prevention previously and received active study agent within 3 months of randomization.
18. Known allergy to ATG or any product excipient
19. Prior treatment with ATG or known allergy to rabbit-derived products or to any product excipient
20. Prior adverse reactions to heparin.
21. Any condition that in the investigator's opinion may adversely affect study participation will be reviewed by the Study Chair to ensure consistency and adjudicate whether or not the subject may compromise the study results
22. Any screening/baseline laboratory result not otherwise stated out of normal reference range and/or medical history that may increase the risk of the subject's participation in this trial.
23. Previously diagnosed with Stage 3 TID according to ADA criteria (see Appendix 3 for Criteria for diagnosis of diabetes)

Ages: 6 Years to 34 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 2 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-12-17 (Actual); Study Completion 2024-12-17 (Actual)

PRIMARY OUTCOMES:
Progression to Stage 3 T1D | 5 years
  The primary outcome is the elapsed time from random treatment assignment to the development of diabetes or time of last contact among those randomized

CONTACTS AND LOCATIONS:
Locations (22):
- United States (20):
  - Children's Hospital of Orange County, Orange, California
  - University of California - San Francisco, San Francisco, California
  - Stanford University, Stanford, California
  - Barbara Davis Center at University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - University of Florida, Gainesville, Florida
  - University of Miami, Miami, Florida
  - University of South Florida Diabetes Center, Tampa, Florida
  - Emory Children's Center, Atlanta, Georgia
  - Indiana University - Riley Hospital for Children, Indianapolis, Indiana
  - Children's Hospital of Iowa, Iowa City, Iowa
  - University of Minnesota, Minneapolis, Minnesota
  - The Children's Mercy Hospital, Kansas City, Missouri
  - Columbia University-Naomi Berrie Diabetes Center, New York, New York
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Prisma Health, Greenville, South Carolina
  - Vanderbilt Eskind Diabetes Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Utah, Salt Lake City, Utah
  - Benaroya Research Institute, Seattle, Washington
- Australia (2):
  - Queensland Children's Hospital, South Brisbane, Queensland
  - Walter and Eliza Hall Institute of Medical Research, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: Yes
Data will be available at the NIDDK Central Repository

REFERENCES:
- See also: TrialNet — http://www.diabetestrialnet.org